CLINICAL TRIAL: NCT00424021
Title: An Open-Label, Long-Term Study of Ambrisentan in Pulmonary Hypertension Subjects Having Completed Myogen Study AMB-220
Brief Title: Phase 2 Extension Study of Ambrisentan in Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMB-220-E
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2012-01-27 (Estimated); Last update posted 2012-01-27 (Estimated); Status verified 2011-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — ambrisentan

INTERVENTIONS:
Drug: ambrisentan — 1, 2.5, 5, and 10 mg ambrisentan given orally once daily
  Other Names: BSF 208075; Letairis; Volibris

SUMMARY:
AMB-220-E is an international, multicenter, open-label study examining the long-term safety of ambrisentan (BSF 208075) in subjects who have previously completed Myogen study NCT00046319, "A Phase II, Randomized, Double-Blind, Dose-Controlled, Dose-Ranging, Multicenter Study of BSF 208075 Evaluating Exercise Capacity in Subjects with Moderate to Severe Pulmonary Arterial Hypertension".

ELIGIBILITY:
Inclusion Criteria:

* Must have completed Visit 14/Week 24 of the NCT00046319 study.
* Women of childbearing potential must have a negative urine pregnancy test at the Screening/Enrollment Visit and agree to use a reliable double barrier method of contraception until study completion and for >=4 weeks following their final study visit.
* Must have completed the Down-titration Period of NCT00046319 prior to enrollment in AMB-220-E and will meet the following additional criteria:
* Subjects with a diagnosis of HIV must have stable disease status at the time of Screening/Enrollment.
* Must be stable on conventional therapy for PAH for >=4 weeks prior to the Screening Visit.

Exclusion Criteria:

* Chronic prostanoid therapy, or other investigational prostacyclin derivative within 4 weeks prior to the Screening Visit.
* Intravenous inotrope use within 2 weeks prior to the Screening Visit.
* Females who are pregnant or breastfeeding.
* Contraindication to treatment with an endothelin receptor antagonist (ERA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2003-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

REFERENCES:
- See also: Pulmonary Hypertension Association — http://www.phassociation.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed Week 24 of NCT00046319 and responded to ambrisentan were eligible for enrollment. Response to ambrisentan treatment was determined by the investigator at Week 24 of NCT00046319 based on improvement in efficacy, acceptable safety profile, and >= 4 weeks of stable, conventional pulmonary arterial hypertension (PAH) therapy.
Pre-assignment Details: No subjects failed screening. Subjects who completed an optional down-titration period at the end of NCT00046319 were re-titrated if their final dose was 5 mg or 10 mg.
Groups:
- 1 mg: The optimized final dose from the open-label period of AMB 220 (given once daily [QD] by oral administration) was used in this study, with further dose refinement at the investigator's discretion.
- 2.5 mg: The optimized final dose from the open-label period of AMB 220 (given QD by oral administration) was used in this study, with further dose refinement at the investigator's discretion.
- 5 mg; 10 mg: The optimized final dose from the open-label period of AMB 220 (given QD by oral administration) was used in this study, with further dose refinement at the investigator's discretion. Subjects who completed an optional down-titration period at the end of AMB 220 were re-titrated if their final dose was 5 or 10 mg.
Period: NCT00046319 Study Period
Arm/Group | 1 mg | 2.5 mg | 5 mg | 10 mg
Started | 16 | 19 | 16 | 13
Completed | 15 | 16 | 15 | 12
Not Completed | 1 | 3 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Sponsor discretion | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: AMB-220-E Study Period
Arm/Group | 1 mg | 2.5 mg | 5 mg | 10 mg
Started | 2 | 7 | 19 | 26
Completed | 1 | 5 | 14 | 16
Not Completed | 1 | 2 | 5 | 10
Not completed — Adverse Event | 1 | 1 | 3 | 7
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 1 mg; 2.5 mg: The optimized final dose from the open-label period of NCT00046319 (given QD by oral administration) was used in this study, with further dose refinement at the investigator's discretion.
- 5 mg; 10 mg: The optimized final dose from the open-label period of NCT00046319 (given QD by oral administration) was used in this study, with further dose refinement at the investigator's discretion. Subjects who completed an optional down-titration period at the end of AMB 220 were re-titrated if their final dose was 5 or 10 mg.
- Total: Total of all reporting groups
Arm/Group | 1 mg | 2.5 mg | 5 mg | 10 mg | Total
Number analyzed (Participants) | 2 | 7 | 19 | 26 | 54
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline represents the beginning of the current extension study (ie, Week 24 of the parent study, NCT00046319).
  years | 54.0 (12.73) | 43.0 (17.18) | 56.7 (13.48) | 49.0 (15.59) | 51.1 (15.33)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline represents the beginning of the current extension study (ie, Week 24 of the parent study, NCT00046319).
  Participants
    Female | 1 | 6 | 17 | 22 | 46
    Male | 1 | 1 | 2 | 4 | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 1 | 5 | 13 | 20 | 39
  Black | 1 | 1 | 1 | 1 | 4
  Asian | 0 | 1 | 2 | 0 | 3
  Hispanic | 0 | 0 | 3 | 5 | 8
Years Pulmonary Arterial Hypertension (PAH) Present [Mean (Standard Deviation); unit: Years] — Baseline represents the beginning of the current extension study (ie, Week 24 of the parent study, NCT00046319).
  Years | 2.0 (0.00) | 4.4 (3.87) | 2.7 (2.91) | 4.8 (4.81) | 3.9 (4.07)
6-minute Walk Distance [Mean (Standard Deviation); unit: Meters] — Baseline represents the beginning of the current extension study (ie, Week 24 of the parent study, NCT00046319). N=24 for the 10-mg group and N=52 for the combined ambrisentan group.
  Meters | 462.0 (132.94) | 400.4 (85.13) | 398.8 (111.56) | 410.7 (93.79) | 406.9 (98.56)
Borg Dyspnea Index [Mean (Standard Deviation); unit: Score] — Baseline represents the beginning of the current extension study (ie, Week 24 of the parent study, NCT00046319). Borg Dyspnea Index, a measure of perceived shortness of breath: 0 units on a scale (none) to 10 units on a scale (maximum breathlessness). N=24 for the 10-mg group and N=52 for the combined ambrisentan group.
  Score | 2.5 (0.71) | 1.6 (1.65) | 2.8 (1.77) | 2.9 (1.81) | 2.7 (1.76)
World Health Organization Class [Number; unit: Participants] — Classes: I) pulmonary hypertension (PH); ordinary physical activity not limited or causes increased dyspnea, fatigue, chest pain, or presyncope. II) PH; ordinary physical activity mildly limited and causes increased dyspnea, fatigue, chest pain, or presyncope; comfortable at rest. III) PH; physical activity markedly limited and less than ordinary physical activity causes increased dyspnea, fatigue, chest pain, or presyncope; comfortable at rest. IV) PH; physical activity causes symptoms; signs of right heart failure; dyspnea/fatigue possibly at rest.
  Participants
    I | 1 | 3 | 0 | 4 | 8
    II | 0 | 3 | 11 | 13 | 27
    III | 1 | 1 | 8 | 9 | 19
Primary Diagnosis [Number; unit: Participants] — Baseline represents the beginning of the current extension study (ie, Week 24 of the parent study, NCT00046319).
  Participants
    Idiopathic Pulmonary Arterial Hypertension | 0 | 5 | 12 | 15 | 32
    Mixed Connective Tissue Disease | 0 | 1 | 1 | 5 | 7
    Systemic Lupus Erythematosus | 0 | 0 | 0 | 2 | 2
    Systemic Sclerosis | 1 | 0 | 2 | 0 | 3
    Overlap Syndrome | 0 | 0 | 0 | 1 | 1
    Anorexigen Use | 0 | 0 | 2 | 2 | 4
    Human immunodeficiency virus (HIV) Infection | 1 | 1 | 0 | 0 | 2
    Other | 0 | 0 | 2 | 1 | 3
Height [Mean (Standard Deviation); unit: Centimeters] — Baseline represents the beginning of the current extension study (ie, Week 24 of the parent study, NCT00046319).
  Centimeters | 169.8 (3.11) | 160.6 (11.84) | 163.1 (8.07) | 164.5 (10.03) | 163.7 (9.42)
Weight [Mean (Standard Deviation); unit: Kilograms] — Baseline represents the beginning of the current extension study (ie, Week 24 of the parent study, NCT00046319).
  Kilograms | 66.0 (8.49) | 68.1 (14.97) | 74.6 (21.32) | 76.1 (17.96) | 74.2 (18.51)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pulmonary Arterial Hypertension (PAH) Who Completed the Phase II NCT00046319 Study and Who Experienced Severe Adverse Events (AEs) During Long-term Ambrisentan Exposure
Description: The number of participants in the AMB-220-E analysis set who experienced AEs (including serious AEs) of severe severity (ie, made it impossible to perform routine activities and the subject may have experienced intolerable discomfort or pain) that began after entering AMB-220-E (treatment-emergent AEs) and that occurred in more than 1 participant are summarized by dose group. The AMB-220-E analysis set consisted of all participants who received at least 1 dose of study drug during the AMB-220-E study.
Time Frame: Week 24 (AMB-220-E baseline) to Week 334
Population: The AMB-220-E population consisted of all subjects who received at least 1 dose of study drug during the AMB-220-E study.
Measure: Number; unit: Participants
Arm/Group | 1 mg | 2.5 mg | 5 mg | 10 mg
Number analyzed (Participants) | 2 | 7 | 19 | 26
Participants
  Abdominal Pain NOS | 0 | 1 | 1 | 0
  Alanine Aminotransferase Increased | 0 | 0 | 0 | 2
  Anaemia NOS | 0 | 1 | 1 | 0
  Angina Pectoris | 0 | 0 | 1 | 1
  Aspartate Aminotransferase Increased | 0 | 0 | 0 | 2
  Gastrointestinal Arteriovenous Malformation | 0 | 0 | 0 | 2
  Gastrointestinal Hemorrhage NOS | 0 | 0 | 0 | 2
  Infection NOS | 0 | 0 | 1 | 1
  Oedema Peripheral | 0 | 0 | 1 | 2
  Ovarian Cyst | 0 | 1 | 0 | 1
  Pulmonary Hypertension NOS Aggravated | 0 | 0 | 0 | 4
  Right Ventricular Failure | 0 | 0 | 1 | 6
  Syncope | 0 | 0 | 0 | 4

2. Secondary Outcome: Baseline Measurement in Exercise Capacity as Measured by the 6-minute Walk Test (6MWT) Distance (Baseline [Week 24])
Description: The 6MWT was conducted according to the American Thoracic Society guidelines (ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med 2002; 166(1):111-117.) Primary efficacy analyses were performed for the AMB-220-E analysis set (all subjects who received at least 1 dose of study drug during the AMB-220-E study).
Time Frame: Week 24 (AMB-220-E baseline)
Population: Primary efficacy analyses were performed for the AMB-220-E analysis set (all subjects who received at least 1 dose of study drug during the AMB-220-E study). Results are presented using the last-observation-carried-forward (LOCF) imputation.
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Combined Ambrisentan Treatment: The optimized final dose from the open-label period of NCT00046319 (1, 2.5, 5, or 10 mg once daily by oral administration) was used in this study, with further dose refinement at the investigator's discretion. The small sample size, nonrandomized dose group assignments, and the potential for dose adjustments precluded meaningful comparisons between the dose groups. Therefore, efficacy results are only presented for the combined ambrisentan group. Results are presented using the LOCF imputation.
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Meters | 406.1 (97.78)

3. Secondary Outcome: Change From Baseline (Week 24 of NCT00046319) in Exercise Capacity as Measured by the 6-minute Walk Test (6MWT) Distance (Last Observation Carried Forward [LOCF]) (Week 48)
Description: as for outcome 2
Time Frame: 24 weeks (Week 24 to Week 48)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Combined Ambrisentan Treatment: The optimized final dose from the open-label period of NCT00046319 (1, 2.5, 5, or 10 mg QD by oral administration) was used in this study, with further dose refinement at the investigator's discretion. The small sample size, nonrandomized dose group assignments, and the potential for dose adjustments precluded meaningful comparisons between the dose groups. Therefore, efficacy results are only presented for the combined ambrisentan group.
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Meters | 4.5 (46.93)
Statistical Analysis 1: Comparison: Combined Ambrisentan Treatment; The small sample size, nonrandomized dose group assignments, and the potential for dose adjustments precluded meaningful comparisons between the dose groups. Therefore, efficacy results are only presented for the combined ambrisentan group; Test type: Superiority or Other; Mean Difference (Net) = 4.5, 95% CI 2-sided [-8.3 to 17.3], Standard Deviation 46.93

4. Secondary Outcome: Change From Baseline (Week 24 of NCT00046319) in Exercise Capacity as Measured by the 6-minute Walk Test (6MWT) Distance (LOCF) (Week 108)
Description: as for outcome 2
Time Frame: 84 weeks (Week 24 to Week 108)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Meters | -10.3 (73.16)
Statistical Analysis 1: Comparison: Combined Ambrisentan Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = -10.3, 95% CI 2-sided [-30.3 to 9.7], Standard Deviation 73.16

5. Secondary Outcome: Change From Baseline (Week 24 of NCT00046319) in Exercise Capacity as Measured by the 6-minute Walk Test (6MWT) Distance (LOCF) (Week 156)
Description: as for outcome 2
Time Frame: 132 weeks (Week 24 to Week 156)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Meters | -4.7 (83.08)
Statistical Analysis 1: Comparison: Combined Ambrisentan Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = -4.7, 95% CI 2-sided [-27.4 to 18.0], Standard Deviation 83.08

6. Secondary Outcome: Change From Baseline (Week 24 of NCT00046319) in Exercise Capacity as Measured by the 6-minute Walk Test (6MWT) Distance (LOCF) (Week 204)
Description: as for outcome 2
Time Frame: 180 weeks (Week 24 to Week 204)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Meters | -13.9 (77.04)
Statistical Analysis 1: Comparison: Combined Ambrisentan Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = -13.9, 95% CI 2-sided [-34.9 to 7.1], Standard Deviation 77.04

7. Secondary Outcome: Baseline Measurement in Exercise Capacity as Measured by the Borg Dyspnea Index (BDI) (Baseline [Week 24])
Description: Change from baseline evaluated after 24 (baseline), 48, 108, 156, and 204 weeks of ambrisentan therapy in BDI (measured as units on a scale) immediately following exercise. Borg Dyspnea Index, a measure of perceived shortness of breath: 0 units on a scale (none) to 10 units on a scale (maximum breathlessness).
Time Frame: Week 24 (AMB-220-E baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Units on a Scale | 2.69 (1.728)

8. Secondary Outcome: Change From Baseline (Week 24 of NCT00046319) in Exercise Capacity as Measured by the BDI (LOCF) (Week 48)
Description: as for outcome 7
Time Frame: 24 weeks (Week 24 to Week 48)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Units on a Scale | 0.21 (1.323)
Statistical Analysis 1: Comparison: Combined Ambrisentan Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = 0.21, 95% CI 2-sided [-0.15 to 0.57], Standard Deviation 1.323

9. Secondary Outcome: Change From Baseline (Week 24 of NCT00046319) in Exercise Capacity as Measured by the BDI (LOCF) (Week 108)
Description: as for outcome 7
Time Frame: 84 weeks (Week 24 to Week 108)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Units on a Scale | 0.46 (1.659)
Statistical Analysis 1: Comparison: Combined Ambrisentan Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = 0.46, 95% CI 2-sided [0.01 to 0.92], Standard Deviation 1.659

10. Secondary Outcome: Change From Baseline (Week 24 of NCT00046319) in Exercise Capacity as Measured by the BDI (LOCF) (Week 156)
Description: as for outcome 7
Time Frame: 132 weeks (Week 24 to Week 156)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Units on a Scale | 0.50 (1.888)
Statistical Analysis 1: Comparison: Combined Ambrisentan Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = 0.50, 95% CI 2-sided [-0.02 to 1.02], Standard Deviation 1.888

11. Secondary Outcome: Change From Baseline (Week 24 of NCT00046319) in Exercise Capacity as Measured by the BDI (LOCF) (Week 204)
Description: as for outcome 7
Time Frame: 180 weeks (Week 24 to Week 204)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Units on a Scale | 0.46 (1.721)
Statistical Analysis 1: Comparison: Combined Ambrisentan Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = 0.46, 95% CI 2-sided [-0.01 to 0.93], Standard Deviation 1.721

12. Secondary Outcome: Baseline Measurement in Exercise Capacity as Measured by the World Health Organization (WHO) Functional Classification (Baseline [Week 24])
Description: Classes: I) pulmonary hypertension (PH); ordinary physical activity not limited or causes increased dyspnea, fatigue, chest pain, or presyncope. II) PH; ordinary physical activity mildly limited and causes increased dyspnea, fatigue, chest pain, or presyncope; comfortable at rest. III) PH; physical activity markedly limited and less than ordinary physical activity causes increased dyspnea, fatigue, chest pain, or presyncope; comfortable at rest. IV) PH; physical activity causes symptoms; signs of right heart failure; dyspnea/fatigue possibly at rest.
Time Frame: Week 24 (AMB-220-E baseline)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Participants
  WHO Classification I | 8
  WHO Classification II | 27
  WHO Classification III | 19
  WHO Classification IV | 0

13. Secondary Outcome: Exercise Capacity as Measured by the WHO Functional Classification (LOCF) After 24 Weeks of Treatment in AMB-220-E
Description: Classes: I) PH; ordinary physical activity not limited or causes increased dyspnea, fatigue, chest pain, or presyncope. II) PH; ordinary physical activity mildly limited and causes increased dyspnea, fatigue, chest pain, or presyncope; comfortable at rest. III) PH; physical activity markedly limited and less than ordinary physical activity causes increased dyspnea, fatigue, chest pain, or presyncope; comfortable at rest. IV) PH; physical activity causes symptoms; signs of right heart failure; dyspnea/fatigue possibly at rest.
Time Frame: 24 weeks (Week 24 [baseline of AMB-220-E] to Week 48)
Measure: Number; unit: Participants
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Participants
  WHO Classification I | 7
  WHO Classification II | 29
  WHO Classification III | 18
  WHO Classification IV | 0

14. Secondary Outcome: Exercise Capacity as Measured by the WHO Functional Classification (LOCF) After 84 Weeks of Treatment in AMB-220-E
Description: as for outcome 13
Time Frame: 84 weeks (Week 24 of NCT00046319 to Week 108)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Participants
  WHO Classification I | 5
  WHO Classification II | 25
  WHO Classification III | 21
  WHO Classification IV | 3

15. Secondary Outcome: Exercise Capacity as Measured by the WHO Functional Classification (LOCF) After 132 Weeks of Treatment in AMB-220-E
Description: as for outcome 13
Time Frame: 132 weeks (Week 24 of NCT00046319 to Week 156)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Participants
  WHO Classification I | 10
  WHO Classification II | 18
  WHO Classification III | 24
  WHO Classification IV | 2

16. Secondary Outcome: Exercise Capacity as Measured by the WHO Functional Classification (LOCF) After 180 Weeks of Treatment in AMB-220-E
Description: as for outcome 13
Time Frame: 180 weeks (Week 24 of NCT00046319 to Week 204)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Participants
  WHO Classification I | 10
  WHO Classification II | 19
  WHO Classification III | 23
  WHO Classification IV | 2

17. Secondary Outcome: Baseline Measurement in Exercise Capacity as Measured by the Subject Global Assessment (SGA) (Baseline [Week 24])
Description: The SGA was determined using a visual-analog scale. Subjects were asked the question, "How are you feeling today?" and were asked to draw a vertical mark on a 100-mm horizontal line in which zero represented "very poor" and 100 represented "excellent."
Time Frame: Week 24 (AMB-220-E baseline)
Population: Primary efficacy analyses were performed for the AMB-220-E analysis set (all subjects who received at least 1 dose of study drug during the AMB-220-E study).
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Units on a Scale | 69.5 (20.49)

18. Secondary Outcome: Change From Baseline (Week 24 of NCT00046319) in Exercise Capacity as Measured by the SGA (LOCF) (Week 48)
Description: as for outcome 17
Time Frame: 24 weeks (Week 24 to Week 48)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Units on a Scale | -0.6 (19.41)
Statistical Analysis 1: Comparison: Combined Ambrisentan Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = -0.6, 95% CI 2-sided [-5.9 to 4.7], Standard Deviation 19.41

19. Secondary Outcome: Change From Baseline (Week 24 of NCT00046319) in Exercise Capacity as Measured by the SGA (LOCF) (Week 108)
Description: as for outcome 17
Time Frame: 84 weeks (Week 24 to Week 108)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Units on a Scale | -7.4 (25.79)
Statistical Analysis 1: Comparison: Combined Ambrisentan Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = -7.4, 95% CI 2-sided [-14.4 to -0.3], Standard Deviation 25.79

20. Secondary Outcome: Change From Baseline (Week 24 of NCT00046319) in Exercise Capacity as Measured by the SGA (LOCF) (Week 156)
Description: as for outcome 17
Time Frame: 132 weeks (Week 24 to Week 156)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Units on a Scale | -5.1 (25.31)
Statistical Analysis 1: Comparison: Combined Ambrisentan Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = -5.1, 95% CI 2-sided [-12.0 to 1.8], Standard Deviation 25.31

21. Secondary Outcome: Change From Baseline (Week 24 of NCT00046319) in Exercise Capacity as Measured by the SGA (LOCF) (Week 204)
Description: as for outcome 17
Time Frame: 180 weeks (Week 24 to Week 204)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 54
Units on a Scale | -1.9 (23.69)
Statistical Analysis 1: Comparison: Combined Ambrisentan Treatment; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = -1.9, 95% CI 2-sided [-8.4 to 4.6], Standard Deviation 23.69

22. Secondary Outcome: Time to Clinical Worsening of PAH
Description: Clinical worsening of PAH was defined as death, lung transplantation, hospitalization for PAH, atrial septostomy, the addition of approved prostanoid therapy, or study withdrawal due to the addition of other clinically approved PAH therapeutic agents. Sildenafil, a type 5 phosphodiesterase (PDE-5) inhibitor, had not received regulatory approval for the treatment of PAH until late in the conduct of AMB 220 and AMB 220-E, and did not count toward clinical worsening. Results are presented as the Kaplan-Meier estimate (% probability) of not having clinical worsening after a given time.
Time Frame: Week 0 (NCT00046319 baseline) to Week 360
Population: The NCT00046319 analysis set (all subjects who received at least 1 dose of study drug during the AMB-220 study) was evaluated during the NCT00046319 and AMB-220-E study periods.
Measure: Number; unit: Probability (%)
Groups:
- Combined Ambrisentan Treatment: The optimized final dose from the open-label period of NCT00046319 (1, 2.5, 5, or 10 mg once daily by oral administration) was used in this study, with further dose refinement at the investigator's discretion. The small sample size, nonrandomized dose group assignments, and the potential for dose adjustments precluded meaningful comparisons between the dose groups. Therefore, efficacy results are only presented for the combined ambrisentan group.
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 64
Probability (%)
  No clinical worsening after 1 year of treatment | 78 (116.662)
  No clinical worsening after 2 years of treatment | 69
  No clinical worsening after 3 years of treatment | 60
  No clinical worsening after 4 years of treatment | 55

23. Secondary Outcome: Failure-free Treatment Status
Description: Failure-free treatment status was defined as the time from initiation of active treatment to the first occurrence of death, lung transplantation, the addition of approved prostanoid therapy, or study withdrawal due to the addition of other clinically approved PAH therapeutic agents. Results are presented as the Kaplan-Meier estimate (% probability) of not having treatment failure after a given time.
Time Frame: Week 0 (NCT00046319 baseline) to Week 360
Population: The NCT00046319 analysis set (all subjects who received at least 1 dose of study drug during the NCT00046319 study) was evaluated during the NCT00046319 and AMB-220-E study periods.
Measure: Number; unit: Probability (%)
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 64
Probability (%)
  No treatment failure after 1 year of treatment | 89 (110.672)
  No treatment failure after 2 years of treatment | 77
  No treatment failure after 3 years of treatment | 74
  No treatment failure after 4 years of treatment | 70

24. Secondary Outcome: Long-term Survival
Description: Long-term survival was defined as the time from initiation of active treatment to death. Results are presented as the Kaplan-Meier estimate (% probability) of survival after a given time.
Time Frame: Week 24 (AMB-220-E baseline) to Week 329.3
Population: The AMB-220-E analysis set (all subjects who received at least 1 dose of study drug during the AMB-220-E study) was evaluated during the AMB-220-E study period.
Measure: Number; unit: Probability (%)
Arm/Group | Combined Ambrisentan Treatment
Number analyzed (Participants) | 64
Probability (%)
  Survival after 1 year of treatment | 94 (111.873)
  Survival after 2 years of treatment | 87
  Survival after 3 years of treatment | 87
  Survival after 4 years of treatment | 87

25. Primary Outcome: Number of Participants With PAH Who Completed the Phase II NCT00046319 Study and Who Experienced AEs of Moderate Severity During Long-term Ambrisentan Exposure
Description: The number of participants in the AMB-220-E analysis set who experienced AEs (including serious AEs) of moderate severity (ie, interfered with routine activities and subject may have experienced significant discomfort) that began after entering AMB-220-E (treatment-emergent AEs) and that occurred in more than 1 participant are summarized by dose group. The AMB-220-E analysis set consisted of all participants who received at least 1 dose of study drug during the AMB-220-E study.
Time Frame: Week 24 (AMB-220-E baseline) to Week 329.3
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- 1 mg: The optimized final dose from the open-label period of NCT00046319 (1, 2.5, 5, or 10 mg QD by oral administration) was used in this study, with further dose refinement at the investigator's discretion.
- 2.5 mg: The optimized final dose from the open-label period of AMB 220 (1, 2.5, 5, or 10 mg QD by oral administration) was used in this study, with further dose refinement at the investigator's discretion.
- 5 mg; 10 mg: The optimized final dose from the open-label period of AMB 220 (1, 2.5, 5, or 10 mg QD by oral administration) was used in this study, with further dose refinement at the investigator's discretion. Subjects who completed an optional down-titration period at the end of AMB 220 were re-titrated if their final dose was 5 or 10 mg.
Arm/Group | 1 mg | 2.5 mg | 5 mg | 10 mg
Number analyzed (Participants) | 2 | 7 | 19 | 26
Participants
  Abdominal Distension | 0 | 1 | 0 | 1
  Activated Partial Thromboplastin Time Prolonged | 0 | 0 | 2 | 0
  Alanine Aminotransferase Increased | 2 | 0 | 0 | 0
  Anaemia NOS | 0 | 0 | 0 | 2
  Angina Pectoris | 1 | 0 | 0 | 1
  Anxiety | 0 | 0 | 1 | 2
  Arthralgia | 1 | 0 | 3 | 5
  Arrhythmia NOS | 0 | 0 | 1 | 1
  Aspartate Aminotransferase Increased | 2 | 0 | 0 | 0
  Atrial Fibrillation | 0 | 0 | 0 | 2
  Back Pain | 0 | 0 | 2 | 2
  Basal Cell Carcinoma | 0 | 0 | 0 | 2
  Bronchitis NOS | 1 | 3 | 1 | 4
  Bronchospasm NOS | 1 | 0 | 0 | 1
  Bursitis | 0 | 0 | 0 | 2
  Calcinosis | 0 | 1 | 1 | 0
  Cataract | 1 | 0 | 0 | 2
  Cellulitis | 0 | 0 | 2 | 0
  Chest Pain | 0 | 3 | 2 | 0
  Constipation | 0 | 0 | 3 | 3
  Contusion | 0 | 0 | 1 | 1
  Cough | 1 | 1 | 2 | 2
  Cyanosis NOS | 0 | 1 | 0 | 1
  Depression | 0 | 0 | 2 | 5
  Diarrhoea NOS | 0 | 0 | 3 | 2
  Dizziness | 0 | 1 | 2 | 2
  Dyspepsia | 0 | 0 | 1 | 1
  Dyspnoea Exacerbated | 0 | 2 | 5 | 1
  Dyspnoea NOS | 0 | 1 | 0 | 2
  Ear Infection NOS | 0 | 0 | 1 | 1
  Epistaxis | 0 | 0 | 0 | 2
  Erythema | 0 | 0 | 1 | 1
  Fatigue | 0 | 0 | 2 | 1
  Fatigue Aggravated | 0 | 0 | 1 | 1
  Flushing | 0 | 1 | 1 | 0
  Foot Fracture | 0 | 0 | 2 | 0
  Gamma-glutamyltransferase Increased | 1 | 0 | 0 | 1
  Gastroenteritis NOS | 0 | 0 | 0 | 2
  Gastroenteritis Viral NOS | 0 | 0 | 1 | 2
  Gastrooesophageal Reflux Disease | 0 | 1 | 1 | 2
  Gingival Infection | 0 | 0 | 1 | 1
  Gout | 0 | 0 | 2 | 0
  Headache | 0 | 0 | 0 | 2
  Hepatobiliary Disorders | 0 | 0 | 1 | 4
  Herpes Zoster | 0 | 0 | 0 | 2
  Hypertension NOS | 0 | 0 | 2 | 0
  Hypokalaemia | 0 | 0 | 1 | 2
  Hypotension NOS | 1 | 0 | 1 | 1
  Hypoxia | 0 | 1 | 1 | 2
  Influenza | 0 | 1 | 1 | 1
  Insomnia | 0 | 0 | 2 | 4
  International Normalised Ratio Increased | 0 | 1 | 2 | 2
  Intervertebral Disc Herniation | 0 | 0 | 1 | 1
  Iron Deficiency Anaemia | 0 | 1 | 1 | 0
  Limb Injury NOS | 0 | 0 | 1 | 1
  Localised Infection | 0 | 0 | 1 | 1
  Localised Osteoarthritis | 0 | 0 | 1 | 1
  Lower Respiratory Tract Infection NOS | 0 | 0 | 0 | 2
  Menorrhagia | 0 | 0 | 0 | 3
  Migraine NOS | 0 | 0 | 0 | 2
  Nasal Congestion | 0 | 0 | 2 | 1
  Nasopharyngitis | 0 | 0 | 1 | 1
  Nausea | 0 | 0 | 1 | 5
  Nausea Postoperative | 0 | 0 | 1 | 2
  Neck Pain | 0 | 0 | 2 | 0
  Oedema Peripheral | 0 | 0 | 1 | 4
  Oesophageal Candidiasis | 0 | 1 | 0 | 1
  Osteoporosis NOS | 0 | 0 | 2 | 0
  Otitis Media NOS | 0 | 0 | 1 | 1
  Pain in Limb | 0 | 0 | 1 | 3
  Palpitations | 0 | 0 | 0 | 2
  Pneumonia NOS | 0 | 0 | 1 | 1
  Post Procedural Pain | 0 | 0 | 0 | 2
  Prothrombin Time Prolonged | 0 | 0 | 2 | 0
  Pruritus | 0 | 0 | 3 | 1
  Pulmonary Hypertension NOS Aggravated | 0 | 1 | 3 | 3
  Pyrexia | 0 | 1 | 0 | 1
  Right Ventricular Failure | 0 | 1 | 1 | 3
  Sinusitis Chronic NOS | 0 | 0 | 0 | 2
  Sinusitis NOS | 0 | 0 | 0 | 5
  Skin Infection | 0 | 0 | 1 | 1
  Syncope | 0 | 1 | 3 | 1
  Tooth Infection | 0 | 1 | 0 | 1
  Tooth Injury | 0 | 1 | 0 | 1
  Upper Respiratory Tract Infection NOS | 1 | 1 | 3 | 8
  Upper Respiratory Tract Infection Viral NOS | 0 | 0 | 0 | 2
  Urinary Tract Infection NOS | 0 | 0 | 4 | 3
  Visual Disturbance NOS | 0 | 1 | 0 | 1
  Vomiting NOS | 0 | 1 | 0 | 1

26. Primary Outcome: Number of Participants With PAH Who Completed the Phase II NCT00046319 Study and Who Experienced AEs of Mild Severity During Long-term Ambrisentan Exposure
Description: The number of participants in the AMB-220-E analysis set who experienced AEs (including serious AEs) of mild severity (ie, did not interfere with routine activities and the subject may have experienced slight discomfort) that began after entering AMB-220-E (treatment-emergent AEs) and that occurred in more than 1 participant are summarized by dose group. The AMB-220-E analysis set consisted of all participants who received at least 1 dose of study drug during the AMB-220-E study.
Time Frame: Week 24 (AMB-220-E baseline) to Week 329.3
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 1 mg | 2.5 mg | 5 mg | 10 mg
Number analyzed (Participants) | 2 | 7 | 19 | 26
Participants
  Abdominal Distension | 0 | 0 | 1 | 3
  Abdominal Pain Upper | 0 | 0 | 2 | 0
  Acquired Hypothyroidism | 0 | 0 | 1 | 1
  Anaemia NOS | 0 | 1 | 1 | 2
  Anorexia | 0 | 0 | 2 | 1
  Anxiety | 0 | 2 | 2 | 1
  Arrhythmia NOS | 0 | 0 | 1 | 1
  Arthralgia | 0 | 2 | 0 | 4
  Asthenia | 0 | 0 | 1 | 1
  Blood Alkaline Phosphatase NOS Increased | 0 | 0 | 1 | 1
  Blood Potassium Decreased | 1 | 1 | 0 | 1
  Bradycardia NOS | 1 | 1 | 0 | 0
  Bronchitis NOS | 0 | 1 | 1 | 1
  Bundle Branch Block Right | 0 | 0 | 2 | 0
  Cardiac Murmur NOS | 0 | 0 | 3 | 2
  Chest Pain | 0 | 1 | 1 | 4
  Clubbing | 0 | 0 | 0 | 2
  Colonic Polyp | 0 | 0 | 1 | 1
  Constipation | 0 | 1 | 1 | 2
  Cough | 0 | 2 | 6 | 6
  Crackles Lung | 0 | 0 | 1 | 3
  Cyanosis NOS | 0 | 0 | 0 | 3
  Depression | 0 | 0 | 1 | 1
  Diarrhoea NOS | 0 | 1 | 4 | 4
  Diverticulum NOS | 0 | 1 | 0 | 1
  Dizziness | 1 | 0 | 3 | 3
  Dizziness Postural | 0 | 1 | 0 | 1
  Dry Mouth | 0 | 0 | 1 | 1
  Dry Skin | 0 | 0 | 2 | 1
  Dyspnoea Exacerbated | 0 | 1 | 3 | 1
  Enanthema | 0 | 0 | 0 | 2
  Epistaxis | 1 | 0 | 4 | 1
  Erythema | 0 | 0 | 3 | 0
  Eye redness | 0 | 0 | 1 | 2
  Fatigue | 0 | 1 | 1 | 1
  Fatigue Aggravated | 0 | 0 | 0 | 4
  Flatulence | 0 | 0 | 1 | 1
  Feeling Cold | 0 | 1 | 1 | 1
  Flushing | 0 | 0 | 2 | 2
  Gastroenteritis NOS | 0 | 0 | 1 | 1
  Gastrointestinal Upset | 0 | 1 | 0 | 1
  Gastrooesophageal Reflux Disease | 1 | 1 | 0 | 0
  Haemorrhoids | 0 | 1 | 0 | 1
  Headache | 1 | 0 | 3 | 6
  Heart Sounds Abnormal | 0 | 1 | 2 | 2
  Hepatomegaly | 0 | 2 | 0 | 2
  Herpes Simplex | 0 | 0 | 0 | 2
  Hypercholesterolaemia | 1 | 0 | 1 | 0
  Hypertension NOS | 0 | 0 | 1 | 2
  Hyperuricaemia | 0 | 1 | 1 | 0
  Hypokalaemia | 1 | 0 | 1 | 1
  Hypotension NOS | 0 | 0 | 3 | 0
  Influenza | 0 | 1 | 0 | 1
  Influenza Like Illness | 0 | 0 | 2 | 0
  Insomnia | 0 | 1 | 1 | 4
  International Normalised Ratio Increased | 0 | 0 | 2 | 0
  Lymphadenopathy | 0 | 0 | 2 | 1
  Muscle Cramp | 0 | 0 | 1 | 1
  Nail Fungal Infection NOS | 0 | 0 | 1 | 1
  Nasal Congestion | 1 | 0 | 4 | 5
  Nasopharyngitis | 0 | 1 | 2 | 5
  Nausea | 0 | 0 | 2 | 5
  Neck Pain | 0 | 0 | 1 | 1
  Nocturia | 0 | 0 | 2 | 0
  Oedema Peripheral | 1 | 3 | 10 | 9
  Oxygen Saturation Decreased | 0 | 0 | 1 | 1
  Pain in Jaw | 0 | 0 | 0 | 2
  Palpitations | 0 | 1 | 3 | 4
  Pericardial Effusion | 0 | 0 | 0 | 2
  Pharyngitis | 1 | 0 | 1 | 3
  Pneumonia NOS | 0 | 0 | 1 | 1
  Productive Cough | 0 | 2 | 0 | 0
  Pruritus | 0 | 0 | 2 | 2
  Pyrexia | 0 | 1 | 3 | 1
  Rash NOS | 0 | 0 | 1 | 3
  Renal Cyst NOS | 0 | 0 | 0 | 2
  Respiratory Tract Infection NOS | 0 | 0 | 1 | 2
  Scleroderma | 0 | 1 | 0 | 1
  Seasonal Allergy | 1 | 0 | 1 | 1
  Sinusitis NOS | 0 | 0 | 1 | 3
  Skin Ulcer | 0 | 0 | 2 | 0
  Sleep Apnoea Syndrome | 0 | 0 | 0 | 2
  Somnolence | 0 | 0 | 1 | 1
  Squamous Cell Carcinoma | 0 | 1 | 0 | 1
  Syncope | 0 | 1 | 2 | 0
  Tachycardia NOS | 0 | 0 | 1 | 2
  Thyroid Disorder | 0 | 0 | 0 | 2
  Transient Ischaemic Attack | 0 | 0 | 0 | 2
  Upper Respiratory Tract Infection NOS | 0 | 3 | 2 | 6
  Vein Distended | 0 | 0 | 1 | 3
  Venous Stasis | 0 | 0 | 0 | 2
  Vertigo | 0 | 0 | 1 | 1
  Viral Infection NOS | 0 | 0 | 1 | 1
  Vision Blurred | 0 | 0 | 1 | 1
  Vomiting NOS | 0 | 1 | 0 | 1
  Weight Decreased | 1 | 0 | 0 | 1
  White Blood Cell Count Increased | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 1 mg | 2.5 mg | 5 mg | 10 mg
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/7 | 12/19 | 18/26
Other Adverse Events (participants affected / at risk) | 2/2 | 7/7 | 19/19 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg (N=2) | 2.5 mg (N=7) | 5 mg (N=19) | 10 mg (N=26)
Anaemia NOS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Secondary anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia NOS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 8 (11)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal symptom NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Inguinal hernia NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction NOS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calcinosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute NOS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal wall infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lobar pneumonia NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function tests NOS abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral arterial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasovagal attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction NOS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension NOS aggravated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous ulcer NOS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg (N=2) | 2.5 mg (N=7) | 5 mg (N=19) | 10 mg (N=26)
Anaemia NOS (Blood and lymphatic system disorders) | 0 (0) | 2 (5) | 2 (5) | 4 (5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukopenia NOS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (1)
Arrhythmia NOS (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Bradycardia NOS (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Clubbing (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cyanosis NOS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Palpitations (Cardiac disorders) | 0 (0) | 1 (2) | 3 (7) | 6 (8)
Palpitations aggravated (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Tachycardia NOS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pigmented naevus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensation of block in ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Acquired hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thyroid disorder NOS (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cataract bilateral NOS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye redness (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual disturbance NOS (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
Abdominal pain NOS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (5) | 5 (8)
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea NOS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 7 (13) | 6 (6)
Diverticulum NOS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Gastrointestinal upset (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (3) | 2 (5)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanosis coli (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4) | 10 (12)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting NOS (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Calcinosis (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 4 (8) | 2 (3) | 4 (5)
Chest pressure sensation (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Enanthema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Fall (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (2) | 3 (5) | 2 (2)
Fatigue aggravated (General disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Lethargy (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal oedema NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 3 (8) | 12 (20) | 15 (26)
Pain NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (3) | 3 (4) | 2 (2)
Rigors (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
Influenza (Infections and infestations) | 0 (0) | 2 (4) | 1 (1) | 2 (3)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (5) | 1 (1)
Nail fungal infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesphageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Otitis media NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia NOS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Respiratory tract infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Respiratory tract infection viral NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 8 (9)
Sinusitis chronic NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin fungal infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory tract infection NOS (Infections and infestations) | 1 (2) | 4 (9) | 5 (7) | 14 (23)
Upper respiratory tract infection viral NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection NOS (Infections and infestations) | 0 (0) | 1 (2) | 4 (10) | 4 (6)
Viral diarrhoea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Abrasion NOS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Limb injury NOS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Nausea postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Open wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Activated partial thromboplastin time (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Blood alkaline phosphatase NOS increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood amylase increased (Investigations) | 1 (4) | 0 (0) | 0 (0) | 1 (1)
Blood chloride decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Cardiac murmur NOS (Investigations) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Carotid bruit (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Heart sounds abnormal (Investigations) | 0 (0) | 1 (4) | 2 (2) | 2 (2)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 4 (7) | 2 (2)
Lipase increased (Investigations) | 1 (4) | 0 (0) | 0 (0) | 1 (1)
Mean cell haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Mean cell volume increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary arterial wedge pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
QRS axis abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous pressure jugular increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Appetite decreased NOS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetes mellitus NOS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 2 (2) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (5) | 9 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc herniation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Knee deformity NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Monoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Muscle cramp (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Osteoarthritis NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pain in limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Polymyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Breast cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Uterine fibroids (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balance impaired NOS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burning sensation NOS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (4) | 5 (9) | 5 (6)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (3) | 3 (3) | 8 (9)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Migraine NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 4 (5) | 3 (5)
Vasovagal attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (4) | 3 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 7 (7)
Depression aggravated (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 8 (11)
Insomnia exacerbated (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cystitis NOS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal cyst NOS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amenorrhoea NOS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast mass NOS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pelvic pain NOS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prostatic hypertrophy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrage (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (7) | 2 (2) | 5 (5)
Bronchospasm NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 3 (5) | 9 (10) | 8 (11)
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (6) | 9 (12) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4) | 3 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 3 (3)
Lung infiltration NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 6 (8) | 6 (7)
Nasal mucosal disorder NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5) | 3 (4) | 6 (13)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (3) | 3 (5)
Productive cough (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pulmonary congestion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension NOS aggravated (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (5) | 7 (8)
Pulmonary vascular disorder NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory fremitus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic NOS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ronchi (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing aggravated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Eczema weeping (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (2)
Hair disorder NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Nail disorder NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (6) | 3 (3)
Rash NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Skin lesion NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Solar keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Sweating increased (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urticaria NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (2) | 3 (3) | 2 (2)
Haematoma NOS (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hot flushes NOS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension NOS (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypotension NOS (Vascular disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (3)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vein distended (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (8)
Venous stasis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Venous ulcer NOS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest tightness (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The small sample size, nonrandomized dose group assignments, and the potential for dose adjustments precluded meaningful comparisons between the dose groups. Therefore, efficacy results are only presented for the combined ambrisentan group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No